CLINICAL TRIAL: NCT02783222
Title: EFFECT: A Randomized Phase II Study to Evaluate the EFficacy and Impact on Function of Two Different Doses of Nab-paclitaxEl in Elderly Patients With advanCed breasT Cancer
Brief Title: EFficacy and Impact on Function of Two Different Doses of Nab-paclitaxEl in Elderly With advanCed breasT Cancer
Acronym: EFFECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Sandro Pitigliani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFECT; 2012-002707-18 (EudraCT Number)
Record Dates: First submitted 2016-04-28; First posted 2016-05-26 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; elderly patients
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B (Active Comparator): Nab-paclitaxel 125 mg/mq weekly for 3 out of every 4 weeks
  Interventions: Drug: Nab-paclitaxel
- Arm A (Experimental): Nab-paclitaxel 100 mg/mq weekly for 3 out of every 4 weeks
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — comparison of different dosages of drug
  Other Names: Abraxane

SUMMARY:
This is a randomized study evaluating the efficacy and impact on function of two different doses of nab-Paclitaxel in elderly patients with advanced breast cancer.

DETAILED DESCRIPTION:
This open-label, randomized phase II trial evaluates in parallel two doses of nab-Paclitaxel (100 and 125mg/m2) given weekly for 3 weeks every 28 days, in elderly women aged 65 years or older, as first line treatment for advanced breast cancer (locally recurrent or metastatic). A short geriatric evaluation of co-morbidity and functional status will be performed before study entry. The functional status will be monitored at baseline and at every cycles during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer, locally recurrent and/or metastatic; any estrogen/progesterone receptor status; HER2 receptor negative OR HER2 positive but with contraindication to anti-HER2 therapy (e.g. known congestive cardiac failure).
* Measurable disease or non-measurable but evaluable disease according to RECIST 1.1 criteria
* ECOG performance status 0-2
* Estimated life expectancy of ≥ 12 weeks
* No known active/symptomatic CNS metastases
* No previous chemotherapy for breast cancer in the advanced setting
* Adequate organ function including ( Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L; Bilirubin ≤ 1.5 mg/dL; ALT and AST ≤ 3 x ULN (with or without known hepatic metastases); ALP ≤ 2.5 x ULN; Serum creatinine ≤ 1.5 ULN or calculated creatinine clearance (CrCl) ≥ 50mL/min according to the Cockcroft Gault formula
* Written informed consent (according to ICH/GCP and national/local regulations)

Exclusion Criteria:

* Significant peripheral neuropathy (significant peripheral neuropathy is defined as ≥ grade 2 on CTCAE v4.0 criteria)
* Clinically significant comorbidities including: uncontrolled cardiac arrhythmias (except rate-controlled atrial fibrillation), NYHA class III or IV cardiac failure, uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity
* Other malignancy within the last 5 years, except for adequately treated non-melanomatous skin cancers, cervical intraepithelial neoplasia or cervical carcinoma in situ
* Intake of any concomitant medications or therapies that may potentially interact with the trial agent. Any prohibited medication must be discontinued at least 14 days prior to trial entry
* Presence of any psychological, familial, sociological or geographical condition that may potentially hamper compliance with the study protocol and follow-up schedule; these conditions should be discussed with the patient before trial registration

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Every 12 weeks, until disease progression or death or trial completion (12 months after randomization of the last patient).
  Event is defined as either disease progression or death, or functional decline. Functional decline is defined as decreased in at least 1 point from baseline ADL, and/or IADL, as confirmed by the investigator as treatment-related and confirmed at the subsequent cycle

SECONDARY OUTCOMES:
Objective response rate (ORR) | Every 12 weeks, until disease progression or trial completion (12 months after randomization of the last patient).
  Documentation of disease response or progression will be based on RECIST 1.1 criteria
Clinical benefit rate (CBR) | Every 12 weeks, until disease progression or trial completion (12 months after randomization of the last patient)
  Documentation of disease response or progression will be based on RECIST 1.1 criteria
Progression free survival (PFS) | Every 12 weeks, until disease progression or death or trial completion (12 months after randomization of the last patient)
  Documentation of disease progression will be based on RECIST 1.1 criteria
Overall survival (OS) | Every 12 weeks until death or trial completion (12 months after randomization of the last patient)
  Documentation of death
Incidence of adverse events | Every 12 weeks until event occurrence or trial completion (12 months after randomization of the last patient)
  Severity will be reported based on CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Laura Biganzoli, MD, Principal Investigator — Azienda USL Toscana Centro - Prato
Locations (14):
- Italy (14):
  - A.O.U. Ospedali Riuniti, Ancona
  - Centro Di Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - Spedali Civili Brescia, Brescia
  - Ospedale Antonio Perrino, Brindisi
  - Ospedale Ss. Trinita', Frosinone
  - Ospedale Vito Fazzi, Lecce
  - Ausl 12 Viareggio, Lucca
  - Istituto Europeo Oncologia, Milan
  - A.O.U. Federico Ii Di Napoli, Napoli
  - Istituto Oncologico Veneto, Padua
  - Fondazione Maugeri, Pavia
  - A.O.U. S. Maria Della Misericordia Di Udine, Udine
  - Ospedale Civile Maggiore, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biganzoli L, Cinieri S, Berardi R, Pedersini R, McCartney A, Minisini AM, Caremoli ER, Spazzapan S, Magnolfi E, Brunello A, Risi E, Palumbo R, Leo S, Colleoni M, Donati S, De Placido S, Orlando L, Pistelli M, Parolin V, Mislang A, Becheri D, Puglisi F, Sanna G, Zafarana E, Boni L, Mottino G. EFFECT: a randomized phase II study of efficacy and impact on function of two doses of nab-paclitaxel as first-line treatment in older women with advanced breast cancer. Breast Cancer Res. 2020 Aug 5;22(1):83. doi: 10.1186/s13058-020-01319-1. PMID 32758299